CLINICAL TRIAL: NCT01955941
Title: Characterization of Vascular Response to Brachytherapy Using Functional Optical Coherence Tomography
Brief Title: Vascular Response to Brachytherapy Using Functional OCT
Status: Completed | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Alison Skalet, Alison Skalet, MD, PhD, Assistant Professor of Ophthalmology, Oregon Health and Science University
Other Study IDs: IRB00009501; IRB#00009501 (Other: OHSU Institutional Review Board)
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Uveal Melanoma
Keywords: Uveal melanoma; brachytherapy; radiation; ciliary body; choroid; I-125 plaque brachytherapy
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort A: Patients with uveal melanoma for which brachytherapy is recommended will be considered and evaluated for enrollment into this study in order to describe the association between radiation treatment and changes in vision and blood flow within these treated eyes. Changes in vision and blood flow will be monitored at yearly intervals over a 5-year period. Up to 60 subjects will be recruited for this group.
- Cohort B: Patients with uveal melanoma who have previously undergone I-125 plaque brachytherapy will be considered for enrollment into this study to evaluate blood flow in eyes with more advanced radiation-induced changes. This group will only undergo a one-time study session. Up to 40 subjects will be recruited for this group.

SUMMARY:
The purpose of this study is to learn how blood flows to tumors in patients treated with I-125 plaque brachytherapy for uveal melanoma.

DETAILED DESCRIPTION:
Despite having excellent local tumor control rates, uveal melanoma remains a life-threatening cancer, and even eye-sparing therapy with radiation treatment often leads to significant loss of vision. Major challenges to providing care to patients with uveal melanoma include the inability to accurately predict long-term vision in an eye treated with radiation, due to a poor understanding of the nature of radiation retinopathy and optic neuropathy. Optical coherence tomography (OCT) is a commonly used ophthalmic imaging modality that provides precise, real-time data in vivo in a non-invasive manner. Our research group has recently developed two novel functional OCT technologies: (1) Doppler OCT to quantitatively measure total retinal flow and (2) OCT angiography technology to map optic nerve head, retinal, and choroidal blood flow with unprecedented accuracy. The investigators believe this technology can be utilized to improve understanding of radiation-induced vascular changes in the optic nerve and retina that cause vision loss in patients treated with radiation, as well as provide a tool to monitor tumor response to treatment.

In this study, the investigators intend to utilize these novel functional OCT technologies to describe the changes over time in optic nerve head and retinal blood flow after I-125 radiation therapy, and to evaluate the relationship between changes in flow and decreased vision. The investigators will also study the association between changes in flow and the total radiation doses received by the optic nerve head and macula, which varies based upon tumor location and size.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and older with uveal melanomas involving the ciliary body and/or the choroid undergoing I-125 plaque brachytherapy.

Exclusion Criteria:

* Inability to give informed consent.
* Inability to maintain stable fixation for OCT imaging
* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant
* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
* Blood pressure > 180/110 (systolic above 180 OR diastolic above 110). If blood pressure is brought below 180/110 by anti-hypertensive treatment, subject can become eligible.
* Women who are pregnant or lactating at the time of enrollment due to unknown safety of fluorescein angiography. Women that become pregnant during the course of the study may remain enrolled; however, flurorescein and ICG angiography will not be performed until they are no longer pregnant or nursing an infant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will measure blood flow changes in 28 patients with uveal melanoma requiring radiation therapy.
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Blood flow pattern changes in uveal melanoma patients after radiation treatment (Cohort A) | 60 months
  The purpose of this study is to learn how blood flows to tumors in important structures of the eye in patients treated with I-125 plaque brachytherapy for uveal melanoma. This will be assessed using Doppler OCT and OCT angiography technologies.
Blood flow pattern changes in uveal melanoma in eyes with more advanced radiation-induced changes (Cohort B) | 1 study session
  Describe changes over time in tumor vascularity and vascular caliber as measured by OCT angiography in eyes that have already undergone I-125 plaque therapy and demonstrate signs of radiation-induced changes.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Skalet, MD, PhD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided